CLINICAL TRIAL: NCT03898050
Title: The Ideal Transcutaneous Cardiac Pacer Pad Position Study
Brief Title: Ideal Pacer Pad Position Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Siamak Moayedi, MD, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HP-00085450
Record Dates: First submitted 2019-03-29; First posted 2019-04-01 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Symptomatic Bradycardia
Keywords: transcutaneous pacer pad; transcutaneous cardiac pacing

STUDY DESIGN:
Intervention Model Description: The study will employ a prospective crossover design in which participants will function as their own controls. It will compare the pacing threshold of the two most common pacer pad placement positions. Pad placement order will be randomized to eliminate carry-over effect.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A-P (Experimental): Anterior - Posterior pad placement
  Interventions: Procedure: transcutaneous cardiac pacing
- A-L (Experimental): Anterior - Lateral pad placement
  Interventions: Procedure: transcutaneous cardiac pacing

INTERVENTIONS:
Procedure: transcutaneous cardiac pacing — transcutaneous cardiac pacing

SUMMARY:
Temporary transcutaneous cardiac pacing is a life-saving procedure in patients with unstable bradycardia. The American Heart Association (AHA) guidelines for the management of unstable bradycardia recommend initiating transcutaneous pacing in patients unresponsive to atropine while addressing the primary cause of the bradycardia. The two most commonly described pacer pad application sites are the anterior-posterior (A-P) position (positive pad placed under the left scapula and negative pad placed on the left anterior lower chest wall) and the anterior-lateral (A-L) position (positive pad placed on the right anterior chest wall and negative pad placed on the left lower axilla). Major resuscitation organization (AHA, European, Australian) guidelines and text books of emergency medicine recommendations for pacer pad placement do not address the issue of which set of positions are preferred. There are no published human studies addressing ideal pacer pad placement. This study's objective is to assess if there is a significant difference in the pacing threshold (mA) between these two pacer pad positions. The study hypothesis is that the anterior-posterior position will require a lower current and cause less involuntary muscle contraction. The investigators plan to enroll volunteer human subjects undergoing elective cardioversion in the electrophysiology laboratory for atrial fibrillation/flutter. After successful cardioversion to a sinus rhythm, each subject will be transcutaneously paced to mechanical capture in both pacer pad positions. Optimal placement will be determined by the pad position with the lowest current required for capture. The conclusions of this study will provide evidence for the optimal choice regarding pacer pad placement, which can be used in future resuscitation guidelines.

DETAILED DESCRIPTION:
Temporary transcutaneous cardiac pacing is a life-saving procedure in patients with unstable bradycardia. The American Heart Association (AHA) guidelines for the management of unstable bradycardia recommend initiating transcutaneous pacing in patients unresponsive to atropine while addressing the primary cause of the bradycardia. The two most commonly described pacer pad application sites are the anterior-posterior (A-P) position (positive pad placed under the left scapula and negative pad placed on the left anterior lower chest wall) and the anterior-lateral (A-L) position (positive pad placed on the right anterior chest wall and negative pad placed on the left lower axilla). Major resuscitation organization (AHA, European, Australian) guidelines and text books of emergency medicine recommendations for pacer pad placement do not address the issue of which set of positions are preferred. There are no published human studies addressing ideal pacer pad placement. This study's objective is to assess if there is a significant difference in the pacing threshold (mA) between these two pacer pad positions. The study hypothesis is that the anterior-posterior position will require a lower current and cause less involuntary muscle contraction. The investigators plan to enroll volunteer human subjects undergoing elective cardioversion in the electrophysiology laboratory for atrial fibrillation/flutter. After successful cardioversion to a sinus rhythm, each subject will be transcutaneously paced to mechanical capture in both pacer pad positions. Optimal placement will be determined by the pad position with the lowest current required for capture. The conclusions of this study will provide evidence for the optimal choice regarding pacer pad placement, which can be used in future resuscitation guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Age >17 years.
* Scheduled for cardioversion of supraventricular dysrhythmia in the electrophysiology lab.
* Full decision-making capacity.
* Fluent in English language.

Exclusion Criteria:

* Age <18 years.
* Unable to provide informed consent for any reason (including altered mental status or hemodynamic instability).
* Prisoner, under custody or ward of state.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
cardiac capture mA | one minute
  minimal current of energy required to achieve cardiac capture

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moayedi S, Patel P, Brady N, Witting M, Dickfeld TL. Anteroposterior pacer pad position is better than anterolateral for transcutaneous cardiac pacing. Resuscitation. 2022 Dec;181:140-146. doi: 10.1016/j.resuscitation.2022.11.009. Epub 2022 Nov 18. PMID 36410605